CLINICAL TRIAL: NCT05801354
Title: Turmeric Gel as Alternative Non-Vital Pulpotomy Medicament in Primary Teeth-A Randomized Controlled Trial
Brief Title: Turmeric Gel as Alternative Non-vital Pulpotomy Medicament in Primary Teeth
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Collaborators: Lahore General Hospital (Other Government)
Responsible Party: Principal Investigator, Dr. Mashal Mazhar, Dental Surgeon (Ex-Postgraduate trainee), University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UHSUniversity
Record Dates: First submitted 2023-02-28; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Non-Vital Tooth
MeSH Terms: conditions — Tooth, Nonvital | interventions — formocresol

STUDY DESIGN:
Intervention Model Description: Turmeric gel= interventional drug Formocresol= Control drug (standard drug)
Who Masked: Participant, Outcomes Assessor
Masking Description: patients and assessors involved in the study from randomization, allocation, bacteriological outcome, and data analysis will be blinded to which medicament group the patients belonged as all data will be coded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Formocresol (Control-Gold standard-Group A) (Active Comparator): Premade Formocresol (Tricresol & Formalin) was used composed of Tricresol 35%, Formaldehyde (40%) 19%, excipient additive 100% (PD, Switzerland, ISO9001/ISO9001_2000/ ISO13485/CE_MARK), (Universal Dental Pvt, Ltd).
  Interventions: Drug: Formocresol
- Turmeric gel (Experimental-Group B) (Experimental): Turmeric gel will be self-prepared at the Institute of Microbiology and Molecular Genetics, Punjab University, Lahore. 2kgs of Turmeric rhizomes were purchased from a local market in Lahore and verified by a taxonomist, Botany Department, Government College University, Lahore (voucher number: GC.Herb.Bot.3693). Approximately 170g powder along with 550ml distilled water will be taken in a Soxhlet extractor for 96 hours and then filtered repeatedly through Whatman No.1 filter paper. The obtained filtrate will then be mixed with 6% Sodium Carboxy-Methyl Cellulose (NaCMC) (Genevex Chem, Hyderabad, India) to form gel. Four Vitamin C grounded tablets (Wilson's Vitamin C, Wilson's Healthcare, Islamabad, Pakistan) and twelve Vitamin E capsules (Evion, Martin Dow pharmaceuticals, Ltd. Karachi, Pak) will then be added in 100g of gel as antioxidants.
  Interventions: Drug: Turmeric Gel

INTERVENTIONS:
Drug: Turmeric Gel — Turmeric gel will be used as non-vital pulpotomy medicament compared with Formocresol (which is gold standard)
  Other Names: Medicaments for non-vital pulpotomy procedure
  Arms: Turmeric gel (Experimental-Group B)
Drug: Formocresol — Formocresol will be used as non-vital pulpotomy medicament (which is gold standard)
  Other Names: Medicaments for non-vital pulpotomy procedure
  Arms: Formocresol (Control-Gold standard-Group A)

SUMMARY:
The purpose of this randomized controlled clinical trial is to use Turmeric gel as non-vital Pulpotomy medicament compared to Formocresol in primary teeth by evaluating its antibacterial effect against Streptococcus mutans and Lactobacillus acidophilus. It is hypothesized that there is no difference in the antibacterial effect of Turmeric gel compared with Formocresol, when used as non-vital Pulpotomy medicaments.

DETAILED DESCRIPTION:
It is a multi-arm parallel Randomized Controlled Trial in which forty patients aged between 4 to 8 years, each containing at-least one non-vital primary molar, will be selected and randomly divided into Group A (Formocresol) and Group B (Turmeric gel). Non-vital Pulpotomy will be performed by removing the coronal necrotic pulp. Sterile paper point will be dipped in the root canals and taken to the laboratory. Cotton pellets soaked in the respective medicaments will be placed over the root canal orifices and filled temporarily. Patients will be recalled after one week. Samples will be again taken, and tooth restored. Comparison between bacterial count at baseline and after one week of treatment will be made and expressed as Colony-Forming Units/ml (CFU/ml).

ELIGIBILITY:
Inclusion Criteria:

1. Cooperation of patients and consent of parents.
2. Patients with ASA classification I and II (mild to moderate systemic disease).
3. Non-traumatic extensively carious hence restorable primary molars.
4. No history of antibiotic use for 2 weeks.
5. Presence of following clinical signs or symptoms suggestive of non-vital tooth such as tenderness on percussion, non-responsive to cold test, periapical/furcal radiolucency, localized gingival/mucosal soreness/ redness/ swelling, and/or slight mobility-grade I.

Exclusion Criteria:

1. History of allergy to anesthetics and latex.
2. Radiographic evidence of pulpal floor opening into the furcation area.
3. More than half of the roots resorbed.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-03-02 (Actual)

PRIMARY OUTCOMES:
Antibacterial effect | 1 week
  Bacterial count of S. mutans and L. acidophilus counted as Colony Forming Units/ml (CFU/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Shazia Naz, BDS, MDS, Study Director — Associate Professor of Operative Dentistry (Supervisor)
Locations (1):
- de' Montmorency College of Dentistry, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No